CLINICAL TRIAL: NCT05160350
Title: Investigation of Probiotic Effect on Seizure Frequency of Adult Patients With Drug-resistant Epilepsy; A Randomized Double-blind Parallel Placebo-controlled Clinical Trial
Brief Title: Probiotic in Treatment of Adult Patients With Drug-resistant Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasim Tabrizi, Associate professor of neurology, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6938
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Epilepsy; Treatment
MeSH Terms: conditions — Epilepsy | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Familact 2 plus (Zist takhmir pharmaceutical company, Iran), one capsule per day
  Interventions: Drug: Probiotic
- Placebo (Placebo Comparator): Similar capsule in shape and size (Zist takhmir pharmaceutical company, Iran), one capsule per day
  Interventions: Drug: Probiotic

INTERVENTIONS:
Drug: Probiotic — Each probiotic capsule contained combination of lactobacillus and Bifidobacterium species.
  Other Names: Placebo

SUMMARY:
This study is a randomized, double-blind parallel group placebo-controlled clinical trial with the aim of investigating the effect of probiotic versus placebo on drug-resistant adult patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

Drug resistant epilepsy

Exclusion Criteria:

* Hypersensitivity to probiotic
* Acute pancreatitis
* Pregnancy
* Breastfeeding
* Being under treatment with corticosteroids
* Being under treatment with antibiotics during 2 months before enrollment
* Need for antibiotic therapy during the study
* Change in anti-seizure medication within the month before enrollment

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change in seizure frequency | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bu Ali Sina Hospital, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: No